CLINICAL TRIAL: NCT00623376
Title: Randomized Double Blind Cross Over Study Assessing the Effect of Cannabiniods on Spasticity in Spinal Cord Injured Persons :A Pilot Study
Brief Title: Randomized Double Blind Cross Over Study for Nabilone in Spasticity in Spinal Cord Injury Persons
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Manitoba (Other)
Collaborators: Valeant Canada Limited (Industry)
Responsible Party: Sepideh Pooyania, University of Manitoba
Other Study IDs: 4940
Record Dates: First submitted 2008-02-14; First posted 2008-02-26 (Estimated); Last update posted 2008-02-26 (Estimated); Status verified 2007-06

CONDITIONS: Spasticity in Spinal Cord Injured Persons

ARMS (2):
- 1 (Active Comparator): first on treatment then on Placebo
  Interventions: Drug: nabilone then placebo
- 2 (Placebo Comparator): first on placebo then on treatment
  Interventions: Drug: placebo then nabilone

INTERVENTIONS:
Drug: nabilone then placebo — The subjects were first on Nabilone, then crossed over to placebo
  Arms: 1
Drug: placebo then nabilone — the subjects were first on placebo then crossed over to nabilone
  Arms: 2

SUMMARY:
Objectives: To determine whether nabilone, a synthetic cannabinoid, alleviates spasticity in people with spinal cord injury (SCI).

Methods: Twelve subjects were enrolled in this double-blind, placebo-controlled, crossover study. They received either nabilone or placebo during the first four-week period (0.5mg OD with option to increase to 0.5mg BID), then outcome measures were assessed. After a two-week washout, subjects were crossed-over to the opposite arm.

The primary outcome was the Ashworth scale for spasticity in the most involved muscle group, chosen by the subject and clinician. The secondary outcomes included Spasm Frequency Scale, Visual Analog Scale, Wartenberg Pendulum Test, sum of the Ashworth Scale in eight muscle groups of each side of the body, and the Clinician's and Subject's Global Impression of Change .

ELIGIBILITY:
Inclusion Criteria:

* Patients with spinal cord injury were eligible for the study if they are 18-65 years old, have C5 (ASIA A-D) and below and the injury occurred greater than 1 year previously. They had to have stable neurological level of injury with moderate spasticity (Ashworth >/= 3) and no cognitive impairments. The spasticity medications needed to be unchanged for at least 30 days before inclusion, and no botulinum toxin injections for > 4 months.

Exclusion Criteria:

They were excluded if they had:

* Heart disease as cannabinoids can reduce heart rate and blood pressure
* History of psychotic disorders, schizophrenia or any active psychological disorder
* Previously documented sensitivity to marijuana or other cannabinoid agents
* Severe liver dysfunction
* Cognitive impairment
* Major illness in another body area
* If they were pregnant or nursing mother
* Had history of drug dependency
* Used smoked cannabis < 30 days before the onset of the study or were unwilling not to smoke during the study; OR
* If they fixed tendon contractures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2007-07; Primary Completion 2007-11 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Ashworth scale in most involved group muscles | 10 weeks

SECONDARY OUTCOMES:
The secondary outcomes included Spasm Frequency Scale, Visual Analog Scale, Wartenberg Pendulum Test, sum of the Ashworth Scale in eight muscle groups of each side of the body, and the Clinician's and Subject's Global Impression of Change . | 10 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Rehabilitation hospital ,800 sherbrook St., Winnipeg, Manitoba, Canada